CLINICAL TRIAL: NCT02268019
Title: A Comparison Between Tourniquet Application and Epinephrine Injection for Hemostasis During Hypospadias Surgery: the Effect on Bleeding and Post-operative Outcome
Brief Title: Hemostasis During Hypospadias Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Farshid Alizadeh, Assistant professors of medical science, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUMS2014
Record Dates: First submitted 2014-09-15; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Hypospadias Repair
Keywords: hypospadias; dehiscence; urethral stricture; side effects
MeSH Terms: conditions — Hypospadias; Urethral Stricture | interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypospadiasis repair (Experimental)
  Interventions: Procedure: tourniquet application; Drug: epinephrine injection

INTERVENTIONS:
Procedure: tourniquet application
Drug: epinephrine injection

SUMMARY:
A comparison between the two hemostatic methods of hypospadias repairing operation, in terms of early and mid-term (up to 6 months) failure rate (wound dehiscence and urethral stricture needing reoperation) between the two groups: Group A) diluted Epinephrine injection, Group B) tourniquet application in children

ELIGIBILITY:
Inclusion Criteria:

- age under 15 Hypospadiasis ( Distal, Midshaft, Proximal)

Exclusion Criteria:

- Bleeding tendency Penoscrotal Hypospadiasis Other method

Max Age: 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Bleeding | During surgery

SECONDARY OUTCOMES:
fistula | after surgery for 6 months

OTHER OUTCOMES:
meatal and neourethral stricture | after surgery for 6 months
wound dehiscence | after surgery for 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan University of Medical science, Isfahan, Isfahan, Iran